CLINICAL TRIAL: NCT06983093
Title: Effects of Rain Stick and Musical Egg on Pain, Fear and Anxiety During Blood Collection in Children Aged 4-6: A Randomized Controlled Trial
Brief Title: Effects of Rain Stick and Musical Egg on Pain, Fear and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Demir Kösem, Assistant Professor, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HakkariOU
Record Dates: First submitted 2025-04-26; First posted 2025-05-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Procedural Pain; Procedural Anxiety; Fear Needles
MeSH Terms: conditions — Pain, Procedural; Iatrophobia

STUDY DESIGN:
Intervention Model Description: Intervention Group-Rainstick Group: The rainstick method will be used as a non-pharmacological application for the children in this group. The rainstick will be given to the children and during the blood collection process, the researcher or parent will turn it up and down to watch the sounds and movements and if they wish, they will be allowed to take the toy with their free hand.
  Intervention Group-Musical Egg Group: The musical egg method will be used as a non-pharmacological application for the children in this group. The musical egg will be given to the children and during the blood collection process, the researcher or parent will turn it up and down to watch the sounds and movements and if they wish, they will be allowed to take the toy with their free hand.
  Control Group: The child will be seated in the intervention chair. No pharmacological or non-pharmacological method will be applied to the children in this group other than the routine blood collection process.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to prevent bias, support will be obtained from an independent statistician. In addition, data will be collected by a nurse who does not know the groups not included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rainstick Group (Experimental): Intervention Group-Rainstick Group: The rainstick method will be used as a non-pharmacological application for children in this group. The rainstick will be given to the children and during the blood collection process, the researcher or parent will turn it up and down and watch the sounds and movements and if they wish, they will be allowed to take the toy with their free hand. The rainstick will be cleaned with alcohol after being used on each child. The blood collection process will be performed by the nurse working in the blood collection unit.
  Interventions: Other: Rain Stick
- Musical Egg Group (Experimental): Intervention Group-Musical Egg Group: The musical egg method will be used as a non-pharmacological application for the children in this group. The children will be given a musical egg and during the blood collection process, the researcher or parent will turn it up and down and watch the sounds and movements and if they want, they will be allowed to take the toy with their free hand. The musical egg will be cleaned with alcohol after it is used on each child. The blood collection process will be done by the nurse working in the blood collection unit.
  Interventions: Other: Musical Egg
- Control Group (No Intervention): The child will be taken to the blood collection room after being informed that the mother or father will be with him/her during the procedure. The child will be seated in the intervention chair. No pharmacological or non-pharmacological method will be applied to the children in this group other than routine blood collection. The blood collection will be performed by the nurse working in the blood collection unit.

INTERVENTIONS:
Other: Rain Stick — The rain stick to be used in the study is a toy made of wood, ranging in length from 20 to 120 cm. It is also a very entertaining musical instrument that imitates the sound of real rain. It is suitable for use by children aged 4 to 6. It has spiral shapes and colorful beads inside. When the rain stick is turned up and down, it produces a perfect rain sound that drizzles and patters. It is also known as a rain sound stick. The visual and auditory nature of the rain stick can distract the child during the blood collection process.
  Arms: Rainstick Group
Other: Musical Egg — The musical egg to be used in the study is a toy made of wood, approximately 6.5-7 cm in size. These wooden shaker eggs are a fun and interesting musical instrument. It is suitable for use by children aged 4-6. It is filled with iron sand and when shaken, it makes a clear sound and adds a unique rhythm to the music. This egg imitates the sound of maracas when shaken. Maracas are a musical instrument that makes a sound when shaken thanks to the parts in its hollow body. It is also known as musical eggs, egg shakers, musical egg maracas, Easter egg percussion instruments. The visual and auditory nature of the musical egg can distract the child during the blood collection process.
  Arms: Musical Egg Group

SUMMARY:
This research will be conducted in a pre-test-post-test parallel group randomized controlled experimental study model to determine the effects of rain stick and musical egg applied during blood collection on pain, fear and anxiety in children aged 4-6.

Research Hypotheses H1: The mean pain scores of the children in the rain stick group are lower than the mean scores of the children in the control group.

H2: The mean fear scores of the children in the rain stick group are lower than the mean scores of the children in the control group.

H3: The mean anxiety scores of the children in the rain stick group are lower than the mean scores of the children in the control group.

H4: The mean pain scores of the children in the musical egg group are lower than the mean scores of the children in the control group.

H5: The mean fear scores of the children in the musical egg group are lower than the mean scores of the children in the control group.

H6: The mean anxiety scores of the children in the musical egg group are lower than the mean scores of the children in the control group.

DETAILED DESCRIPTION:
Blood collection is one of the most frequently performed invasive procedures in the health sector for years, and it is a stressful situation for all age groups. It causes intense pain, fear and anxiety, especially for children. Although it is known as the preschool period, especially between the ages of four and under, children believe that the needle puncture procedure will disrupt their body integrity and cause disability, and they think that they are being punished for not listening to their parents. These thoughts can also cause the child to experience pain, fear and anxiety. Negative experiences and pain resulting from invasive procedures can lead to negative situations such as needle phobia and avoidance of healthcare personnel. For all these reasons, invasive procedures, which are an important source of pain, fear and anxiety in children, need to be managed effectively. During painful and stressful medical procedures applied to the child, using a timely and effective method to control pain, fear and anxiety will increase tolerance to pain, fear and anxiety in later applications. Pain, fear and anxiety management requires the work of a multidisciplinary team (nurse, physician, other healthcare personnel). In eliminating children's fear of medical procedures, all healthcare professionals, especially nurses, have important responsibilities as the first people to greet children in the hospital and spend the most time with them. Diagnosing, evaluating, and observing the child's pain, fear, and anxiety, preventing complications by applying non-pharmacological nursing interventions, and administering analgesics upon doctor's request are among the roles and responsibilities of nurses. Nurses involved in the treatment of pain, fear, and anxiety carry out a complex care process by applying medical and complementary treatments together. In particular, non-pharmacological complementary treatments, which are independent nursing roles, are effectively applied in eliminating pain, fear, and anxiety symptoms. Various studies emphasize the importance of nursing interventions in preventing and reducing pain, fear and anxiety in children during invasive procedures and controlling the negativities that will be reflected in the treatment process. One of the most frequently preferred non-pharmacological methods for controlling pain, fear, and anxiety that occur during invasive procedures in children is distraction. This method is a nursing intervention that allows the patient's attention to be better controlled by focusing the pain and anxiety elsewhere. With this method, the child protects himself from feeling pain. Distraction methods can be helpful in reducing children's perception of pain, increasing pain tolerance, and providing relaxation, especially during invasive procedures. There are many different methods used to distract attention. Some of these are; listening to music, playing games, using distraction cards, watching cartoons, blowing balloons, creating balloons by blowing foam, watching kaleidoscopes and using virtual reality glasses. In order for distraction methods to be effective, they must be appropriate for the child's age. In the preschool period, audio and visual toys can be effective in distracting children's attention. Play is a tool that helps the child's ability to cope with and adapt to problems by transferring their experiences and fears related to traumatic events that disturb their self to play and toys, and thus reducing pain, fear and anxiety. It is reported that during play, the child's handling and familiarization with the tools used in treatment will reduce pain, fear and anxiety by perceiving them as less threatening. In a study, it was observed that a lighted rotating musical toy used as one of the techniques to divert attention during the blood collection process of preschool children (4-6 age group) reduced the children's pain and fear levels. When the studies in the literature were examined, it was seen that there were limited studies examining the effect of a lighted, moving, musical toy on pain and anxiety in children between the ages of 4-6 during the blood collection procedure in that age group. In this case, it is difficult for nurses to decide on the practices they will use based on the limited research results regarding the use of musical toys in children during blood collection procedures. In the literature review, no studies were found investigating the effects of musical toys such as rain sticks and musical eggs on pain, fear, and anxiety in children during blood collection procedures. Therefore, it is thought that this randomized controlled and experimental study will contribute to the literature and nurses in the field, and will be useful in terms of creating an evidence-based resource for nursing science.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 4-6 years old
* The child must not have acute pain
* The child must not have mental or auditory disabilities
* The child must not have confusion
* The child and parent must agree to participate in the study

Exclusion Criteria:

* The child must be under 4 years old and over 6 years old
* The child's body temperature must be 38°C or above
* The child must have used an analgesic medication in the last 24 hours before the application

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain During Blood Collection Procedure in Children | "1 year"
  It is an unpleasant, emotional and sensory feeling that originates from any part of the body, is accompanied by real or potential tissue damage, and encompasses all past experiences of the patient.
Fear During Blood Collection Procedure in Children | "1 year"
  It is a vital reaction that occurs as a stimulus response as a result of a specific pain or an event perceived as a threat.
Anxiety During Blood Collection Procedure in Children | "1 year"
  It is a psychiatric disorder that causes intense anxiety and worry about possible future threats that are perceived but not present.

IPD SHARING:
Plan to Share IPD: No